## Blood Biomarkers for diagnosis and prognosis of concussion

**CONSENT FORM** 

NCT NUMBER: NCTXXXXXXXXX

08/MAY/2019

## Study Title: Blood Biomarkers for diagnosis and prognosis of concussion

| Subject Number: | | |
|---|---|---|
| Principal Investigator: Dr John Mulvihill | | |
| Participation in this study is voluntary and you may withdra | aw at any time for any i | reason |
| | Please tick app | ropriate box |
| The research project and procedure associated with it have been fully explained to me. | YES | NO |
| All experimental procedures have been identified and no guarantees have been given about the possible results. | YES | NO |
| I have had the opportunity to ask questions concerning any and all aspects of the project and any procedures involved. | YES | NO |
| I am aware that participation is voluntary and I may withdraw consent at any time. | YES | NO |
| I am aware that my decision not to participate or to withdraw will not restrict my access to health care services normally available to me. | YES | NO |
| Confidentiality of records concerning my involvement in this project will be maintained in an appropriate manner and my data is protected. | YES | NO |
| I understand that portions of my team medical records may be looked at by responsible individuals from the research team. I give permission for these individuals to have access to my records. | YES | NO |
| I understand that the investigators have such insurance as is required by law in the event of injury resulting from this research | YES | NO |
| Analyses of all samples and information collected will be conducte<br>some occasions the analyses may be done in collaboration with<br>partners, which may require samples to be shipped to and/or ana<br>cases, samples and data will be coded with anonymized identifier no | third parties, including co<br>lysed by these organisation | ommercial |
| I am happy that the samples and data will be stored and used in ot topic of research (i.e. neurological disorders). | ther research studies within its withing the research studies within its window its within its window its wind | n this |
| Page 1 of 2 | Land Don II you agree) | |

ICF Concussion Study Version 5.0  $8^{\text{th}}$  May 2019

## Study Title: Blood Biomarkers for diagnosis and prognosis of concussion

| Access to my samples and/or my data will require approval fr | om the L | Ехеси | tive Mana | ngement | Group of |
|---|---|---|---|---|---|
| the Faculty of Science and Engineering, University of Limerick. | | | | | |
| (ple | ase tick | box | if you a | gree) | |
| Any identified biomarkers from this study can be used and dis | seminate | d by | the princi | ipal inve | stigator. |
| (ple | ase tick | box | if you a | gree) | |
| I agree that my contact details may be made available for a fo | • | | • | | lowing my |
| participation in this project or its Clinical Research Ethics Committee approved collaborators. | | | | | |
| (plea | ase tick | box i | if you ag | ree) | |
| I, the undersigned, hereby consent to participate as a subject in University of Limerick. I have received a copy of this consent for leaflet for my records. I understand that if I have any question Dr. John Mulvihill, Biomedical Engineer, University of L | orm and a | a copy<br>ning t | of the pa | atient in | formation |
| Telephone number: (061) 237719. | | | | | |
| Subject's Signature: | Date: | | | | - |
| | | dd | mon | уу | |
| NAME (BLOCK LETTERS): | Time: | | | | _ |
| Dagagashaw'a Ciroak wa | Data | | | | |
| Researcher's Signature: | Date: | dd | mon | уу | - |
| NAME (BLOCK LETTERS) | Time | | | | |
| TWITE (DEOCK LETTERO) | i ii i i c. | | | | - |

Page 2 of 2